CLINICAL TRIAL: NCT05437861
Title: Return to Work - Will Brief Intervention Reduce Opioid-induced Back Pain? A RCT Pilot Study
Brief Title: Return to Work - Will Brief Intervention Reduce Opioid-induced Back Pain?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Akershus (Other)
Collaborators: Et liv i bevegelse (ELIB) (Unknown)
Responsible Party: Principal Investigator, Johannes Gjerstad, Project manager, University Hospital, Akershus
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 21/08211
Record Dates: First submitted 2022-05-30; First posted 2022-06-29 (Actual); Last update posted 2022-06-29 (Actual); Status verified 2022-06

CONDITIONS: Opioid Dependence; Low Back Pain; Opioid Use
MeSH Terms: conditions — Opioid-Related Disorders; Low Back Pain | interventions — Crisis Intervention

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment as usual (No Intervention)
- Brief Intervention (Experimental)
  Interventions: Behavioral: Brief Intervention

INTERVENTIONS:
Behavioral: Brief Intervention — A short conversation with the participant regarding their use of opioids will be conducted. During the conversation the participants potential drug dependency will be uncovered. Further the pros and cons of weaning of the medication will be explained and a new treatment plan will be proposed.
  Arms: Brief Intervention

SUMMARY:
Background Back pain is among the most common cause for sick leave in the working population and is the main cause of years lived with disability globally. In Norway, about 30% report to live with chronic pain and women are affected more than men. Pharmacological strategies for pain management e.g., opioid medications, is a common treatment method. This is despite clinical guidelines suggesting limiting pharmacological treatment in management of chronic back pain. Long-term use of opioids is linked to opioid-induced hyperalgesia, paradoxically. However, it is suggested that RNA sequencing (seq.) profiling may identify individuals that are at risk of opioid-induced hyperalgesia. To help reduce medication intake brief intervention (BI), a method for discontinuing long-term medication use, has shown to be successful. In this pilot RCT the investigators aim to investigate the feasibility of a full scale RCT and observational study using BI on opioid-using patients with back pain and concurrently study if the response can be predicted by RNA seq.

Method Ten outpatients aged 18-67 years with back pain will be recruited from the orthopaedic department at Akershus University Hospital. Inclusion criteria includes daily use of opioids for more than two weeks consecutively, and sufficient language (Norwegian) skills. Exclusion criteria includes severe medical or surgical condition such as cauda equina syndrome, rheumatic disease, psychiatric disease, or recent surgery. The patients will be randomised into two groups (5+5) where one group receives the BI and the other gets treatment as usual. Data collection will be conducted at three-time points; baseline, four weeks follow-up and three months follow-up (end of trial). The primary outcome for this pilot RCT is to test feasibility and estimate effect size for a later full-scale study. Secondary outcomes include subjective and objective findings from the data collection.

Results Primary results concerning feasibility are mainly qualitative and will be presented as such. Secondary results including demographic information as well as tentative effect size, patient reported outcomes such as pain intensity, anxiety, depression, quality of life, psychosocial stressors in the workplace and the RNA seq will be presented descriptively.

Conclusion The results from this pilot study will assist in constructing the optimal design for a full-scale RCT.

ELIGIBILITY:
Inclusion Criteria:

* age 18-67 years, admitted from their GP to Ahus due to back pain,
* daily use of opioids such as ≥ 30 mg codeine or ≥ 45 mg tramadol or ≥ 3 mg oxycodone or other opioids corresponding to a morphine equivalent dose ≥ 10-20 mg

Exclusion Criteria:

* cauda equina syndrome
* recent surgery (within 1 month)
* pregnancy
* psychiatric disease
* rheumatic disease
* diabetic polyneuropathy
* cancer
* insufficient proficiency in the Norwegian language
* no remaining work potential and/or permanent sick pension.

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-08 (Estimated); Primary Completion 2023-01 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the study protocol | 4 months
  Feasibility of the pilot study protocol will be defined as absence of premature discontinuation of treatment. Semi structured interviews will be conducted to collect the therapists and the participants experience in relation to strengths and weaknesses of the protocol. This will help optimize the design for a full scale study. Also questions will be added pertaining to the participants experience of the intervention. This will be uncovered through a conversation at the end of the study.
Power and sample size calculations | 4 months
  Estimate the appropriate sample size for a full-scale study. This will be conducted utilizing a 2-sample t-test

SECONDARY OUTCOMES:
Hopkins symptom check list (HSCL-25) | baseline, 1 month and 4 months
  Assess for changes in questionnaire response regarding change in mental distress, anxiety and/or depression between the 3 time points and feasibility of use of questionnaire battery. Higher score means worse outcome. 4-point likert scale with 25 items.
Gene expression analysis | baseline and 1 month
  This analysis explores gene expression levels from blood samples. The investigaters collect blood samples which are prepared and shipped to the United Kingdom for RNA sequencing. This is conducted by the commercial company Novogene, UK. For updated information about tools and equipment used for RNA sequencing please confer with the company's website (https://en.novogene.com/)
Severity of dependence scale | baseline, 1 month and 4 months
  Assess for changes in medication dependence by investigating questionnaire response between the 3 time points and feasibility of use of questionnaire battery. Higher score means worse outcome.
Questions about substance abuse (DSM-IV) | baseline, 1 month and 4 months
  Assess for changes in medication use by investigating questionnaire response between the 3 time points and feasibility of use of questionnaire battery. Higher score means worse outcome.
Teppers abusive supervision scale | baseline, 1 month and 4 months
  Assess for changes in questionnaire response between the 3 time points and feasibility of use of questionnaire battery. Higher score means worse outcome. 5 items on a 5 point likert scale.
Health related quality of life (EuroQoL 5D) | baseline, 1 month and 4 months
  Assess for changes in health related quality of life by investigating questionnaire response between the 3 time points and feasibility of use of questionnaire battery. Higher score means better outcome.
Visual analogue scale | baseline, 1 month and 4 months
  Assess for changes in reported pain levels by investigating questionnaire response between the 3 time points and feasibility of use of questionnaire battery. Higher score means worse outcome. Score 0-10.